CLINICAL TRIAL: NCT03611725
Title: Comparison of Success Rate Between Distal Radial Approach and Radial Approach in ST-segment Elevation Myocardial Infarction
Brief Title: Comparison of Success Rate Between Distal Radial Approach and Radial Approach in STEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: Hanmi Pharmaceutical co., ltd. (Other)
Responsible Party: Principal Investigator, Seung Hwan Lee, Professor, Wonju Severance Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRAMI
Record Dates: First submitted 2018-07-17; First posted 2018-08-02 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Distal Radial Artery Approach; ST Elevation Myocardial Infarction
Keywords: Distal radial approach; ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Patients will be randomized either distal radial approach or radial approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Distal radial artery (Active Comparator): After subcutaneous injection of lidocaine, the distal radial artery around the bony surface area is punctured with a 20-gauge venipuncture catheter needle or steel needle according to the operator's discretion. After successful puncture, flexible, straight plastic 0.025" mini-guidewire is inserted through the hole of the puncture needle. Then, Radifocus® introducer sheath (Terumo, Tokyo, Japan) is inserted into the distal radial artery.
  Interventions: Procedure: Distal radial artery
- Radial artery (Placebo Comparator): After subcutaneous injection of lidocaine, the radial artery is punctured with a 20-gauge venipuncture catheter needle or steel needle according to the operator's discretion. After successful puncture, flexible, straight plastic 0.025" mini-guidewire is inserted through the hole of the puncture needle. Then, Radifocus® introducer sheath (Terumo, Tokyo, Japan) is inserted into the radial artery.
  Interventions: Procedure: Radial artery

INTERVENTIONS:
Procedure: Distal radial artery — The distal radial artery will be punctured with a puncture needle. Then, coronary angiography and percutaneous coronary intervention will be performed.
  Arms: Distal radial artery
Procedure: Radial artery — The radial artery will be punctured with a puncture needle. Then, coronary angiography and percutaneous coronary intervention will be performed.
  Arms: Radial artery

SUMMARY:
ST-segment elevation myocardial infarction (STEMI) is an emergent disease to treat as soon as possible. 2017 ESC guidelines for the management of STEMI recommend using radial approach (RA) rather than femoral approach (FA) to reduce mortality and bleeding complications if the operators are expert for RA. Recently, Ferdinand Kiemeneij reported that distal radial approach (DRA) could be a feasible and safe route for coronary angiography (CAG) and percutaneous coronary intervention (PCI) in 70 patients. The right-handed patient could feel more comfortable in left DRA than right RA. Left DRA also could provide a better comfortable position for the operator compared to left RA. Distal radial artery is located around the anatomical snuffbox, which doesn't contain nerve and vein beside artery. Therefore, the possibility of procedure-related complications such as nerve injury or arteriovenous fistula is very low. Also, the superficial location of DRA could make easier hemostasis. There were no vascular-related complications from the report of Kiemeneij. But, the rate of puncture failure was 11%, which was higher than RA-based study (5.34% in STEMI patients of RIVAL trial, 6% in RIFLESTEACS trial and 5.8% in MATRIX trial). Nevertheless, this study was a pilot study with a small number of patients. There is no clinical study to compare the feasibility and safety for CAG and PCI between DRA and RA in patients with STEMI. Therefore, this study aimed to evaluate whether DRA is feasible and safe compared to RA in STEMI setting.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* ST-segment elevation myocardial infarction
* Palpable unilateral distal radial and radial artery

Exclusion Criteria:

* Cardiogenic shock
* Thrombolysis before primary percutaneous coronary intervention
* Inability to obtain written informed consent
* Patient with ipsilateral arteriovenous fistula
* Participation in another ongoing clinical trial
* Pregnancy
* Expected lifespan <12 months

  * Eligible operator criteria
* Qualified operator who had experienced ≥ 100 cases of distal radial artery puncture

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Puncture success rate (%) | Through procedure completion, up to 6 hours
  The success rate (%) of arterial puncture will be compared between distal radial artery approach and radial artery approach group.

SECONDARY OUTCOMES:
Success rate of coronary angiography (%) | Through procedure completion, up to 6 hours
  The success rate (%) of coronary angiography will be compared between distal radial artery approach and radial artery approach group.
Success rate of percutaneous coronary intervention (%) | Through procedure completion, up to 6 hours
  The success rate (%) of percutaneous coronary intervention will be compared between distal radial artery approach and radial artery approach group.
Procedure success rate (%) | Through procedure completion, up to 6 hours
  The success rate (%) of final procedure will be compared between distal radial artery approach and radial artery approach group.
Bleeding complication rate (%) | During hospitalization, up to 1 month
  The bleeding complication rate (%) will be compared between distal radial artery approach and radial artery approach group.
Total procedure time (minutes) | Through procedure completion, up to 6 hours
  Scale range: 0 - 360 minutes Shorter time is associated with better outcome. An averaged time value will be compared and reported between two groups.
Total fluoroscopic time (minute) | Through procedure completion, up to 6 hours
  Scale range: 0 - 360 minutes Shorter time is associated with better outcome. An averaged time value will be compared and reported between two groups.
Total fluoroscopic dose (Gray/cm2) | Through procedure completion, up to 6 hours
  Scale range: 0 - 500 Gray/cm2 Lesser fluoroscopic dose is better. An averaged value will be compared and reported between two groups.
MACE (%) | 1 month
  Incidence rate (%) of composite endpoints defined as all-cause death, any myocardial infarction, and any revascularization
Puncture time (minute) | Through procedure completion, up to 6 hours
  Scale range: 0 - 60 minutes Shorter time is considered better result. An averaged time value will be compared and reported between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hwan Lee, MD, Principal Investigator — Yonsei University Wonju College of Medicine, Wonju Severance Christian Hospital
Locations (3):
- South Korea (3):
  - Kangwon National University College of Medicine, Chuncheon, Gangwon-do
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - The Catholic university of Korea Uijeongbu St. Mary's hospital, Uijeongbu-si, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JW, Kim CJ, Lee BK, Ahn SG, Youn YJ, Lee JH, Jeon HS, Kim SY, Jang J, Bu S, Ahn HS, Lim S, Yim HW, Lee SH. Distal Radial Access vs Transradial Access in Patients With ST-Segment Elevation Myocardial Infarction: The DRAMI Trial. JACC Adv. 2025 Nov;4(11 Pt 1):102200. doi: 10.1016/j.jacadv.2025.102200. Epub 2025 Sep 29. PMID 41027079